CLINICAL TRIAL: NCT02276755
Title: Vitamin D in TB Prevention in School Age Children
Brief Title: Vitamin D Supplementation in TB Prevention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Ganmaa Davaasambuu, Assistant Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 140513
Record Dates: First submitted 2014-10-23; First posted 2014-10-28 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Latent Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention: 1 (Active Comparator): Dietary Supplement: Cholecalciferol (vitamin D3)
  Interventions: Dietary Supplement: Cholecalciferol (vitamin D3)
- Placebo Comparator: 2 (Placebo Comparator): Dietary Supplement: Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (vitamin D3) — 14000 IU vitamin D3 weekly Experimental group will receive vitamin D supplement (Tishcon, USA).
  Arms: Intervention: 1
Other: Placebo — Placebo group will receive placebo (Tishcon, USA) weekly.
  Arms: Placebo Comparator: 2

SUMMARY:
The goal of this clinical trial is to determine whether vitamin D supplementation reduces risk of acquiring latent tuberculosis infection (LTBI) in school age children in Mongolia. The investigators hypothesize that (1) vitamin D supplementation will reduce risk of acquisition of LTBI, (2) vitamin D supplementation will safely reduce risk of developing active TB and improve other secondary efficacy outcomes, and (3) children with the lowest vitamin D status at baseline will gain most from the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Boys or girls aged 6 to 13 years at enrolment
2. Attending participating school in Ulaanbaatar at enrolment
3. Child gives informed assent to participate in the study
4. Child's parent/legal guardian gives informed consent for child to participate in study

Exclusion Criteria:

1. Chronic medical conditions
2. Presence of LTBI on screening, as evidenced by a positive QFT-G
3. Clinical signs of rickets, or diagnosis of any other condition requiring vitamin D supplementation
4. Known primary hyperparathyroidism or sarcoidosis
5. Taking immunosuppressant or cytotoxic therapy, or vitamin D supplement > 400IU / day
6. Plans to move away from study area within 3 years of enrolment

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8851 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Acquisition of latent tuberculosis infection | Three years
  The proportion of children who acquire LTBI during the 3 year period will be compared for children randomized to vitamin D3 vs. placebo using the Mantel-Haenszel risk ratio, stratified by school of attendance. The primary analysis will compare the proportion of children who are QuantiFERON-positive at the 0.35 IU/ml IFN-gamma threshold at the end of the study. Exploratory analyses will compare the proportion of children who are positive at the 4.0 IU/ml IFN-gamma threshold (denoting stable conversion) and mean / median antigen-stimulated IFN-gamma concentration analyzed as a continuous variable.

SECONDARY OUTCOMES:
Incidence of active TB disease | Three years
  All participants
Incidence of self-reported acute respiratory infection (upper, lower and both combined) | Three years
  All participants
Incidence of acute respiratory infection requiring hospitalization | Three years
  All participants
Incidence of acute respiratory infections requiring antibiotic treatment | Three years
  All participants
Number of days off school (total number and number due to acute respiratory infection) | Three years
  All participants
Incidence of acute asthma exacerbation requiring hospitalization | Three years
  Sub-set of participants with asthma at baseline
Incidence of new asthma, allergic rhinitis and atopic dermatitis | Three years
  Sub-sets of participants without asthma, allergic rhinitis or atopic dermatitis at baseline
Control of asthma, allergic rhinitis and atopic dermatitis | Three years
  Sub-sets of participants identified as having asthma, allergic rhinitis or atopic dermatitis at baseline
Incidence of bone fracture | Three years
  All participants
Anthropometric outcomes (z-scores for height-for-age, weight-for-age, weight-for-height, body mass index-for-age, and waist circumference and waist-to-height ratio) | Three years
  All participants
Body composition: impedance, impedance%, fat mass fat %, and fat-free mass | Three years
  All participants
Muscle strength: grip strength and long jump distance from standing | Three years
  All participants
Serum 25-hydroxyvitamin D concentration | Three years
  All participants
Bone mineral density at the radius | Three years
  Sub-set of participants
Physical fitness (maximal oxygen consumption estimated from 20m shuttle run) | Three years
  Sub-set of participants
Attention-related behavior scores (Connors III) | Three years
  Sub-set of participants
Incidence of dental caries | Three years
  Sub-set of participants
Circulating and antigen-stimulated concentrations of cytokines, chemokines and other inflammatory mediators | Three years
  Sub-set of participants
Exam performance | Three years
  Sub-set of participants
Self-reported pubertal development | Three years
  Sub-set of participants
Spirometric lung volumes (FEV1 and FVC) | Three years
  Sub-set of participants
Urinary metabolome profile | Three years
  Sub-set of participants
Gut microbiome profile | Three years
  Sub-set of participants

OTHER OUTCOMES:
Incidence of adverse events | Three years
  The proportion of participants experiencing death, one or more serious adverse events of any cause or one or more potential adverse reactions (hypercalcemia, hypercalciuria and hypervitaminosis D) will be compared between arms.
Heterogeneity of treatment effect among sub-groups defined by baseline vitamin D status, estimated calcium intake and vitamin D pathway genotype | Three years
  Heterogeneity of treatment effect will be examined among sub-groups defined by baseline vitamin D status, estimated calcium intake and vitamin D pathway genotype for primary and secondary outcomes. This will be done by repeating efficacy analyses to include:
  1. An interaction term between baseline vitamin D status and allocation to vitamin D vs. placebo
  2. An interaction term between estimated calcium intake and allocation to vitamin D vs. placebo
  3. An interaction term between vitamin D pathway genotype and allocation to vitamin D vs. placebo.
  For genetic analyses, DNA will be extracted from participants' stored whole blood, and typed for a panel of candidate single nucleotide polymorphisms (SNPs) in genes influencing vitamin D metabolism (e.g. CYP2R1, CYP27B1, CYP24A1), transport (e.g. DBP) and signalling (e.g. VDR).
Cost-effectiveness of vitamin D supplementation for the prevention of LTBI and active TB | Three years
  Health economic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Davaasambuu Ganmaa, MD PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Mongolian Health Initiative, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared for purposes of meta-analysis, subject to approval from IRBs in Mongolia and the USA and terms of data sharing agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The items above will be shared following publication of trial reports.
Access Criteria: IPD requests should be made to the Principal Investigator: gdavaasa@hsph.harvard.edu

REFERENCES:
- [Derived] Ganmaa D, Hemmings S, Jolliffe DA, Buyanjargal U, Garmaa G, Adiya U, Tumurbaatar T, Dorjnamjil K, Tserenkhuu E, Erdenenbaatar S, Tsendjav E, Enkhamgalan N, Achtai CE, Talhaasuren Y, Byambasuren T, Ganbaatar E, Purevdorj E, Martineau AR. Influence of vitamin D supplementation on muscle strength and exercise capacity in Mongolian schoolchildren: secondary outcomes from a randomised controlled trial. BMJ Open Sport Exerc Med. 2024 Sep 26;10(3):e002018. doi: 10.1136/bmjsem-2024-002018. eCollection 2024. PMID 39345833
- [Derived] Ganmaa D, Khudyakov P, Buyanjargal U, Tserenkhuu E, Erdenenbaatar S, Achtai CE, Yansanjav N, Delgererekh B, Ankhbat M, Tsendjav E, Ochirbat B, Jargalsaikhan B, Enkhmaa D, Martineau AR. Vitamin D supplements for fracture prevention in schoolchildren in Mongolia: analysis of secondary outcomes from a multicentre, double-blind, randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2024 Jan;12(1):29-38. doi: 10.1016/S2213-8587(23)00317-0. Epub 2023 Dec 1. PMID 38048799
- [Derived] Ganmaa D, Bromage S, Khudyakov P, Erdenenbaatar S, Delgererekh B, Martineau AR. Influence of Vitamin D Supplementation on Growth, Body Composition, and Pubertal Development Among School-aged Children in an Area With a High Prevalence of Vitamin D Deficiency: A Randomized Clinical Trial. JAMA Pediatr. 2023 Jan 1;177(1):32-41. doi: 10.1001/jamapediatrics.2022.4581. PMID 36441522
- [Derived] Ganmaa D, Uyanga B, Zhou X, Gantsetseg G, Delgerekh B, Enkhmaa D, Khulan D, Ariunzaya S, Sumiya E, Bolortuya B, Yanjmaa J, Enkhtsetseg T, Munkhzaya A, Tunsag M, Khudyakov P, Seddon JA, Marais BJ, Batbayar O, Erdenetuya G, Amarsaikhan B, Spiegelman D, Tsolmon J, Martineau AR. Vitamin D Supplements for Prevention of Tuberculosis Infection and Disease. N Engl J Med. 2020 Jul 23;383(4):359-368. doi: 10.1056/NEJMoa1915176. PMID 32706534

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT02276755/Prot_SAP_000.pdf